CLINICAL TRIAL: NCT01072786
Title: A Phase 1 Evaluation of the Safety and Immunogenicity of Five Admixtures of TetraVax-DV, a Recombinant Live Attenuated Tetravalent Dengue Virus Vaccine, in Healthy Flavivirus-naïve Adult Subjects
Brief Title: Evaluation of the Safety and Immune Response of Five Admixtures of a Tetravalent Dengue Virus Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CIR 268
Record Dates: First submitted 2010-02-19; First posted 2010-02-22 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Dengue
Keywords: Dengue Virus; Dengue Fever; Dengue Vaccine; Dengue Hemorrhagic Fever; Dengue Shock Syndrome
MeSH Terms: conditions — Dengue; Severe Dengue

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- TetraVax-DV Vaccine-Admixture 1 (Experimental): Participants will receive the TetraVax-DV admixture 1 vaccine.
  Interventions: Biological: TetraVax-DV Vaccine-Admixture 1
- TetraVax-DV Vaccine-Admixture 2 (Experimental): Participants will receive the TetraVax-DV admixture 2 vaccine.
  Interventions: Biological: TetraVax-DV Vaccine-Admixture 2
- TetraVax-DV Vaccine-Admixture 3 (Experimental): Participants will receive the TetraVax-DV admixture 3 vaccine.
  Interventions: Biological: TetraVax-DV Vaccine-Admixture 3
- TetraVax-DV Vaccine-Admixture 4 (Experimental): Participants will receive the TetraVax-DV admixture 4 vaccine.
  Interventions: Biological: TetraVax-DV Vaccine-Admixture 4
- Placebo (Placebo Comparator): Participants will receive the placebo.
  Interventions: Biological: Placebo
- TetraVax-DV Vaccine-Admixture 5 (Experimental): Participants will receive the TetraVax-DV admixture 5 vaccine.
  Interventions: Biological: TetraVax-DV Vaccine-Admixture 5

INTERVENTIONS:
Biological: TetraVax-DV Vaccine-Admixture 1 — One subcutaneous injection of a recombinant live attenuated TetraVax-DV vaccine, admixture 1 (10^3 PFU of rDEN1Δ30, 10^3 PFU of rDEN2/4Δ30[ME], 10^3 PFU of rDEN3-3´D4Δ30, 10^3 PFU of rDEN4Δ30)
  Arms: TetraVax-DV Vaccine-Admixture 1
Biological: TetraVax-DV Vaccine-Admixture 2 — One subcutaneous injection of a recombinant live attenuated TetraVax-DV vaccine, admixture 2 (10^3 PFU of rDEN1Δ30, 10^3 PFU of rDEN2/4Δ30[ME], 10^3 PFU of rDEN3-3´D4Δ30, 10^3 PFU of rDEN4Δ30-200,201)
  Arms: TetraVax-DV Vaccine-Admixture 2
Biological: TetraVax-DV Vaccine-Admixture 3 — One subcutaneous injection of a recombinant live attenuated TetraVax-DV vaccine, admixture 3 (10^3 PFU of rDEN1Δ30, 10^3 PFU of rDEN2/4Δ30[ME], 10^3 PFU of rDEN3Δ30/31-7164, 10^3 PFU of rDEN4Δ30)
  Arms: TetraVax-DV Vaccine-Admixture 3
Biological: TetraVax-DV Vaccine-Admixture 4 — One subcutaneous injection of a recombinant live attenuated TetraVax-DV vaccine, admixture 4 (10^3 PFU of rDEN1Δ30, 10^3 PFU of rDEN2/4Δ30[ME], 10^3 PFU of rDEN3Δ30/31-7164, 10^3 PFU of rDEN4Δ30-200,201)
  Arms: TetraVax-DV Vaccine-Admixture 4
Biological: Placebo — One subcutaneous injection of a placebo containing vaccine diluent but no actual vaccine
  Arms: Placebo
Biological: TetraVax-DV Vaccine-Admixture 5 — One subcutaneous injection of a recombinant live attenuated TetraVax-DV vaccine, admixture 5 (10^3 PFU of rDEN1Δ30, 10^4 PFU of rDEN2/4Δ30(ME), 10^3 PFU of rDEN3Δ30/31-7164, and 10^3 PFU of rDEN4Δ30)
  Arms: TetraVax-DV Vaccine-Admixture 5

SUMMARY:
Dengue viruses can cause dengue fever and other serious health conditions, primarily affecting people living in tropical regions of the world. This study will evaluate the safety and immune responses of five formulations of a tetravalent dengue virus vaccine in healthy adults.

DETAILED DESCRIPTION:
Dengue viruses cause dengue fever and the more severe condition, dengue hemorrhagic fever/shock syndrome. Dengue viruses are common in most tropical and subtropical regions of the world and infection with dengue viruses is the leading cause of hospitalization and death in children in many tropical Asian countries. For these reasons, the World Health Organization (WHO) has made the development of a dengue virus vaccine a top priority. This study will evaluate the safety and immunogenicity of five versions of a live, attenuated, tetravalent dengue virus vaccine called TetraVax-DV.

This study will enroll healthy adults 18-50 years old. Participants will be randomly assigned to receive one of the five versions of TetraVax-DV or placebo. At the vaccination study visit, participants will undergo a medical history review, physical examination, blood and urine collection, and vital sign measurements. Participants will then receive one injection of their assigned vaccine or placebo in the upper arm. After receiving the vaccine, participants will remain in the clinic for 30 minutes for observation. At home, participants will monitor and record their temperature three times a day for 16 days. Additional study visits will occur at Days 2, 4, 6, 8, 10, 12, 14, 16, 21, 28, 42, and 180 for physical exams, assessment of symptoms, and blood and urine collection. Some participants will attend an additional study visit at Day 60.

Participants who received one of the five versions of the vaccine will be asked to take part in an optional substudy that will evaluate the safety and immunogenicity of a second vaccination 6 months after the first vaccination. In the substudy, participants will be randomly assigned to receive either the same vaccine they received in the first part of the study or a placebo vaccine. For 6 months following the second vaccination, participants will attend study visits and take part in the same study procedures that occurred in the first part of the study.

ELIGIBILITY:
Inclusion Criteria:

* In good general health, as determined by physical examination, laboratory screening, and review of medical history
* Available for the duration of the study, approximately 26 weeks post-vaccination
* Willing to participate in the study as evidenced by signing the informed consent document
* Female participants of childbearing potential must be willing to use effective contraception for the duration of the trial. More information on this criterion can be found in the protocol.

Exclusion Criteria:

* Pregnant or breastfeeding
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies
* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the person's ability to understand and cooperate with the requirements of the study
* Screening laboratory values of Grade 1 or above for absolute neutrophil count (ANC), alanine aminotransferase (ALT), and serum creatinine, as defined in the protocol
* Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a person participating in the study or would render the person unable to comply with the study
* Any significant alcohol or drug abuse in the 12 months before study entry which has caused medical, occupational, or family problems, as indicated by medical history
* History of a severe allergic reaction or anaphylaxis
* Severe asthma (emergency room visit or hospitalization in the 6 months before study entry)
* HIV infection, by screening and confirmatory assays
* Hepatitis C virus (HCV) infection, by screening and confirmatory assays
* Hepatitis B virus (HBV) infection, by Hepatitis B surface antigen (HBsAg) screening
* Any known immunodeficiency syndrome
* Use of anticoagulant medications
* Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 42 days prior to or following vaccination; immunosuppressive dose of corticosteroids is defined as 10 mg or more of prednisone equivalent per day for 14 days or longer
* Receipt of a live vaccine within 28 days or a killed vaccine within the 14 days prior to vaccination or anticipated receipt of any vaccine during the 42 days following vaccination
* Absence of spleen
* Receipt of blood products in the 6 months before study entry, including transfusions or immunoglobulin or anticipated receipt of any blood products or immunoglobulin during the 42 days following vaccination
* History or serologic evidence of previous dengue virus infection or other flavivirus infection (e.g., yellow fever virus, St. Louis encephalitis, West Nile virus)
* Previous receipt of a flavivirus vaccine (licensed or experimental)
* Anticipated receipt of any investigational agent in the 42 days before or after vaccination
* Has definite plans to travel to a dengue endemic area during the study
* Refusal to allow storage of specimens for future research

Inclusion Criteria for Substudy:

* Receipt of vaccine at first vaccination
* In good general health, as determined by physical examination and review of medical history
* Available for the duration of the study, approximately 6 months post-vaccination
* Willing to participate in the study as evidenced by signing the informed consent document
* Female participants of childbearing potential must be willing to use effective contraception for the duration of the trial. More information on this criterion can be found in the protocol.

Exclusion Criteria for Substudy:

* Pregnant or breastfeeding
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies
* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the person's ability to understand and cooperate with the requirements of the study
* Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a person participating in the study or would render the person unable to comply with the study
* Any significant alcohol or drug abuse in the past 12 months which has caused medical, occupational, or family problems, as indicated by medical history
* History of a severe allergic reaction or anaphylaxis
* Severe asthma (emergency room visit or hospitalization within the last 6 months)
* HIV infection, by screening and confirmatory assays
* Hepatitis C virus (HCV) infection, by screening and confirmatory assays
* Hepatitis B virus (HBV) infection, by Hepatitis B surface antigen (HBsAg) screening
* Any known immunodeficiency syndrome
* Use of anticoagulant medications
* Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 42 days prior to or following vaccination; immunosuppressive dose of corticosteroids is defined as 10 mg or more of prednisone equivalent per day for 14 days or longer
* Receipt of a live vaccine within 28 days or a killed vaccine within the 14 days prior to vaccination or anticipated receipt of any vaccine during the 42 days following vaccination
* Absence of spleen
* Receipt of blood products within the past 6 months, including transfusions or immunoglobulin or anticipated receipt of any blood products or immunoglobulin during the 42 days following vaccination
* Anticipated receipt of any other investigational agent in the 42 days before or after vaccination
* Has definite plans to travel to a dengue endemic area during the study
* Refusal to allow storage of specimens for future research

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 141 (Actual)
Dates: Start 2010-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Safety of five TetraVax-DV admixtures, as assessed by the frequency of vaccine-related adverse events (AEs), graded by severity | Measured out to Day 28
Determination of the serum plaque reduction neutralization titer 60% (PRNT_60) to DEN1, DEN2, DEN3, and DEN4 viruses | Measured at Days 0, 28, 42, and 180
Monovalent, bivalent, trivalent, and tetravalent seropositivity and seroconversion rates | Measured at 4 and 6 weeks after vaccination
Seropositivity and seroconversion rates to greater than 60% in in the TetraVax-DV admixture 5 vaccine arm | Measured by Day 42

SECONDARY OUTCOMES:
Frequency, quantity, and duration of viremia following vaccination | Measured out to Day 21
Number of vaccinees infected with DEN1, DEN2, DEN3, and DEN4 | Measured by Day 42
Duration of the neutralizing antibody response | Measured at Day 180
Safety and immunogenicity of a second dose of vaccine given 6 months after the first dose (optional substudy) | Measured at Day 222 (42 days after second dose)
Seroconversion as assessed by a greater than or equal to 4-fold rise in DEN1, DEN2, DEN3, or DEN4 neutralizing antibody titers compared with the pre-vaccination antibody titer | Measured by Day 42
Seropositivity as assessed by PRNT_60 to DEN1, DEN2, DEN3, DEN4 greater than or equal to 1:10 compared with the pre-vaccination titer | Measured by Day 42

CONTACTS AND LOCATIONS:
Overall Officials: Anna Durbin, MD, Principal Investigator — Center for Immunization Research (CIR), Johns Hopkins School of Public Health
Locations (4):
- United States (4):
  - Center for Immunization Research, Johns Hopkins School of Public Health, Washington D.C., District of Columbia
  - Center for Immunization Research, Johns Hopkins School of Public Health, Baltimore, Maryland
  - Fletcher Allen Health Care (FAHC), General Clinical Research Center (GCRC), Burlington, Vermont
  - University of Vermont Vaccine Testing Center, Burlington, Vermont

REFERENCES:
- [Background] Durbin AP, McArthur J, Marron JA, Blaney JE Jr, Thumar B, Wanionek K, Murphy BR, Whitehead SS. The live attenuated dengue serotype 1 vaccine rDEN1Delta30 is safe and highly immunogenic in healthy adult volunteers. Hum Vaccin. 2006 Jul-Aug;2(4):167-73. doi: 10.4161/hv.2.4.2944. Epub 2006 Jul 24. PMID 17012875
- [Background] Blaney JE Jr, Durbin AP, Murphy BR, Whitehead SS. Targeted mutagenesis as a rational approach to dengue virus vaccine development. Curr Top Microbiol Immunol. 2010;338:145-58. doi: 10.1007/978-3-642-02215-9_11. PMID 19802584
- [Background] Durbin AP, McArthur JH, Marron JA, Blaney JE, Thumar B, Wanionek K, Murphy BR, Whitehead SS. rDEN2/4Delta30(ME), a live attenuated chimeric dengue serotype 2 vaccine is safe and highly immunogenic in healthy dengue-naive adults. Hum Vaccin. 2006 Nov-Dec;2(6):255-60. doi: 10.4161/hv.2.6.3494. Epub 2006 Nov 5. PMID 17106267
- [Background] Durbin AP, Whitehead SS, McArthur J, Perreault JR, Blaney JE Jr, Thumar B, Murphy BR, Karron RA. rDEN4delta30, a live attenuated dengue virus type 4 vaccine candidate, is safe, immunogenic, and highly infectious in healthy adult volunteers. J Infect Dis. 2005 Mar 1;191(5):710-8. doi: 10.1086/427780. Epub 2005 Jan 27. PMID 15688284
- [Background] McArthur JH, Durbin AP, Marron JA, Wanionek KA, Thumar B, Pierro DJ, Schmidt AC, Blaney JE Jr, Murphy BR, Whitehead SS. Phase I clinical evaluation of rDEN4Delta30-200,201: a live attenuated dengue 4 vaccine candidate designed for decreased hepatotoxicity. Am J Trop Med Hyg. 2008 Nov;79(5):678-84. PMID 18981503
- [Derived] Kirkpatrick BD, Durbin AP, Pierce KK, Carmolli MP, Tibery CM, Grier PL, Hynes N, Diehl SA, Elwood D, Jarvis AP, Sabundayo BP, Lyon CE, Larsson CJ, Jo M, Lovchik JM, Luke CJ, Walsh MC, Fraser EA, Subbarao K, Whitehead SS. Robust and Balanced Immune Responses to All 4 Dengue Virus Serotypes Following Administration of a Single Dose of a Live Attenuated Tetravalent Dengue Vaccine to Healthy, Flavivirus-Naive Adults. J Infect Dis. 2015 Sep 1;212(5):702-10. doi: 10.1093/infdis/jiv082. Epub 2015 Mar 22. PMID 25801652
- [Derived] Durbin AP, Kirkpatrick BD, Pierce KK, Elwood D, Larsson CJ, Lindow JC, Tibery C, Sabundayo BP, Shaffer D, Talaat KR, Hynes NA, Wanionek K, Carmolli MP, Luke CJ, Murphy BR, Subbarao K, Whitehead SS. A single dose of any of four different live attenuated tetravalent dengue vaccines is safe and immunogenic in flavivirus-naive adults: a randomized, double-blind clinical trial. J Infect Dis. 2013 Mar 15;207(6):957-65. doi: 10.1093/infdis/jis936. Epub 2013 Jan 17. PMID 23329850